CLINICAL TRIAL: NCT05822583
Title: Strategies and Treatments for Respiratory Infections &Amp; Viral Emergencies (STRIVE): Immune Modulation Strategy Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STRIVE
Record Dates: First submitted 2023-02-04; First posted 2023-04-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- active treatment group (Experimental): Active treatment group (IV abatacept infusion, 10 mg/kg up to 1750 mg) + baseline IM
  Interventions: Drug: abatacept infusion
- Control group (Placebo Comparator): Placebo group (IV infusion of normal saline) + baseline IM
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: abatacept infusion — The dose of abatacept will be 10 mg/kg given as a single infusion on Day 0, with a maximum dose of 1,750 mg, so any participant with weight of >175 kg will receive a dose of 1750 mg. + baseline IM (immune modulator)
  Arms: active treatment group
Drug: Placebo group — Placebo group (IV infusion of normal saline) + baseline IM
  Arms: Control group

SUMMARY:
COVID-19 can trigger a dysregulated immune response, and previous studies have shown that immune modulation can improve outcomes in hospitalized patients. This trial is designed to determine whether intensification of immune modulation early in the course of the disease (while patients are on low flow oxygen) with abatacept (active arm) combined with standard of care (SOC) improves recovery as compared with placebo + SOC (placebo arm). For both groups, intensification of immunomodulation will be provided as part of SOC in case of signs of disease progression (patient requires high flow nasal oxygen (HFNO) or more support) and/or if the patient has rapidly increasing oxygen requirement.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of SARS-CoV2 infection by nucleic acid test (NAT) or equivalent non-NAT test [list of approved tests in the PIM] within 14 days of randomization.
* Requiring hospitalization for the management of COVID-19
* Has evidence of COVID-19 pneumonia (PNA) defined as either receiving supplementary oxygen ≤2L of low flow oxygen with evidence of airspace disease on chest imaging (X ray, computer tomography or ultrasound) OR receiving supplementary oxygen >2L and <10 L of low flow oxygen.
* Currently receiving or planned to receive (ordered) one IM drug (for example, a corticosteroid or baricitinib) as part of treatment of COVID-19 prior to randomization.
* Has started supplemental oxygen for the treatment of COVID-19 within the past 5 calendar days. Patients on home oxygen are eligible if current oxygen flow rate is increased from baseline and other above criteria are met.
* Investigator agrees that the pneumonia is due to COVID-19.

Exclusion Criteria:

* Oxygen requirement of ≥10L or more of low flow oxygen (or equivalent if using Venturi mask, etc), or requiring either HFNO, NIV, IMV, or ECMO.
* Participant has received more than one baseline IM for treatment of the current COVID-19 infection at time of trial enrollment. (Examples: corticosteroid, baricitinib, tocilizumab, anakinra, abatacept, or infliximab.)
* Participant anticipated to not meet all inclusion criteria within 24 hours of randomization in the opinion of the investigator.
* Allergy to investigational agent.
* Neutropenia (absolute neutrophil count <1000 cells/μL) (<1.0 x 10 3 /μL or <1.0 G/L) on most recent lab within 2 calendar days of randomization.
* Lymphopenia (absolute lymphocyte count <200 cells/μL) (<0.20 x 10 3 /μL or <0.20 G/L) on most recent lab within 2 calendar days of randomization.
* Known or suspected active or recent serious infection (bacterial, fungal, viral, or parasitic infection, excepting SARS-CoV-2) that in the opinion of the investigator could constitute a risk when taking investigational agent. Note: Broad spectrum empiric antibiotic usage does not exclude participation.
* Known or suspected history of untreated tuberculosis (TB). TB diagnosis may be suspected based on medical history and concomitant therapies that would suggest TB infection. Participants are also excluded if they have known, latent TB treated for less than 4 weeks with appropriate anti-tuberculosis therapy per local guidelines (by history only, no screening required).
* Have received any live vaccine (or live attenuated) within 3 months before screening or intend to receive a live vaccine (or live attenuated) during the trial. Use of prior non-live (inactivated) vaccinations is allowed for all participants, including any vaccine for COVID-19.
* Pre-existing immunomodulation or immunosuppression that meets any of the following: Participant has received abatacept for an indication other than COVID- 19 within 5 half-lives (65 days) of enrollment (Abatacept elimination half-life is 13.1 days.) Participant is receiving immune modulatory therapy for autoimmune, transplant management or another indication AND has one or more of the following: evidence of active infection (other than COVID-19) or has required reduction in their immune modulatory therapy in the preceding 6 months due to infectious complication (routine reduction as SOC is not an exclusion) or has required intensification in immunotherapy within the preceding 6 months due to organ rejection/worsening underlying disease status (e.g., intensification with an additional agent on top of usual immunosuppressive regimen)
* Participant has recently received or is anticipated to require immune modulatory agents for their underlying disease including chemotherapeutic treatments likely to induce neutropenia (<1.0 x 10 9 cells/µL) or lymphopenia (<1.0 x 10 9 cells/µL)
* Participant has untreated advanced HIV (known CD4 <200 in the past 6 months) AND is not established on antiretroviral therapy
* Pregnancy
* Breastfeeding
* Co-enrollment in other trials not predetermined to be compatible with this trial.
* In the investigator's judgment, the patient has any advanced organ dysfunction that would not make participation appropriate.
* The treating clinician expects inability to participate in trial procedures or participation would not be in the best interests of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Days to Recovery Scale | 60 days post-intervention
  DRS-60 is a version of the STRIVE clinical recovery scale (CRS) which combines time to recovery with non-recovered clinical state and death to an ordinal outcome.0 indicates best results, 60 represents recovered on Day 60, with not recovered by Day 60 coded as 61 and death (worst outcome) as 62.

SECONDARY OUTCOMES:
time to sustained recovery though Day 60 | baseline to day 60
  Time to sustained recovery is defined as being discharged from the index hospitalization, followed by being alive and home for 14 consecutive days prior to the end of follow-up
all-cause mortality though Day 60 | baseline to day 60
  substantial attempts will be made to determine vital status through the end of follow-up by a combined approach of follow-up visits with the participant or proxy, chart review, and review of other available information sources.
time to progression | baseline to day 60
  will be defined by the study day on which a participant experiences a definite progression.
  Definite progression is defined as a participant requiring HFNO, NIV, IMV, or ECMO therapy, OR, if HFNO is unavailable, a participant requiring ≥15 L/min conventional oxygen.
  Probable progression is defined as a participant not meeting criteria for definite progression but requiring ≥10 L/min conventional oxygen, OR, a participant with an oxygen requirement that has increased by ≥4 L/min in the preceding 24 hours.
Three-category ordinal outcome | Day 60
  assessed at Day 60, with categories "recovered (alive and at home at Day 60)", "alive and not recovered", and dead
the pulmonary ordinal outcome | Day 5, 14, and 28
  categories defined as:
  1. Can independently undertake usual activities with minimal or no symptoms
  2. Symptomatic and currently unable to independently undertake usual activities but no need of supplemental oxygen (or not above premorbid requirements)
  3. Supplemental oxygen <4 liters/min (or <4 liters/min above premorbid requirements)
  4. Supplemental oxygen ≥4 liters/min (or ≥4 liters/min above premorbid requirements, but not high-flow oxygen)
  5. Non-invasive ventilation or high-flow oxygen
  6. Invasive ventilation, extracorporeal membrane oxygenation (ECMO), mechanical circulatory support, or new receipt of renal replacement therapy
  7. Death

CONTACTS AND LOCATIONS:
Overall Officials: Cavan Reilly, PhD, Principal Investigator — University of Minnesota; Christina Barkauskas, MD, Study Chair — Duke University
Locations (127):
- United States (82):
  - University of Alabama Birmingham University Hospital (Site 213-002), Birmingham, Alabama
  - Banner University Medical Center Tucson (Site 206-004), Tucson, Arizona
  - Southern Arizona VA Healthcare System (Site 074-009), Tucson, Arizona
  - UC Davis Health (Site 203-004), Davis, California
  - UCSF Fresno (Site 203-005), Fresno, California
  - VA Loma Linda Healthcare System (074-017), Loma Linda, California
  - MemorialCare Health System (066-003), Long Beach, California
  - VA Long Beach Healthcare System (074-026), Long Beach, California
  - Cedars-Sinai Medical Center (208-002), Los Angeles, California
  - Ronald Reagan UCLA Medical Center (Site 203-002), Los Angeles, California
  - VA Northern California Health Care System (Site 074-023), Mather, California
  - VA San Diego Healthcare System (074-016), San Diego, California
  - Zuckerberg San Francisco General Hospital and Trauma Center (213-007), San Francisco, California
  - UCSF Medical Center at Mount Zion (203-007), San Francisco, California
  - San Francisco VAMC (Site 074-002), San Francisco, California
  - UCSF Medical Center (Site 203-001), San Francisco, California
  - Stanford University Hospital & Clinics (Site 203-003), Stanford, California
  - Rocky Mountain Regional VA Medical Center (Site 074-010), Aurora, Colorado
  - University of Colorado Hospital (Site 204-001), Aurora, Colorado
  - Public Health Institute at Denver Health (Site 017-004), Denver, Colorado
  - Yale University (Site 025-001), New Haven, Connecticut
  - MedStar Health Research Institute (Site 009-021), Washington D.C., District of Columbia
  - Washington DC VA Medical Center (Site 009-004), Washington D.C., District of Columbia
  - Tampa General Hospital (032-001), Tampa, Florida
  - Emory Grady (Site 301-032), Atlanta, Georgia
  - Hope Clinic, Emory University (Site 301-031), Decatur, Georgia
  - University of Illinois at Chicago (008-012), Chicago, Illinois
  - Lutheran Medical Group (301-010), Fort Wayne, Indiana
  - University of Kansas Medical Center (Site 080-044), Kansas City, Kansas
  - Massachusetts General Hospital (202-002), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (202-001), Boston, Massachusetts
  - Lahey Hospital and Medical Center (Site 213-001), Burlington, Massachusetts
  - Baystate Medical Center (Site 201-001), Springfield, Massachusetts
  - University of Massachusetts Chan Medical School (080-007), Worcester, Massachusetts
  - VA Ann Arbor Healthcare System (Site 074-028), Ann Arbor, Michigan
  - University of Michigan Medical Center (205-001), Ann Arbor, Michigan
  - Henry Ford Health System (014-001), Detroit, Michigan
  - Sinai-Grace Hospital (Site 205-005), Detroit, Michigan
  - M Health Fairview University of Minnesota Medical Center (112-001), Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center (Site 202-005), Jackson, Mississippi
  - Washington University School of Medicine (Site 003-001), St Louis, Missouri
  - University of Nebraska Medical Center (Site 080-045), Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center (301-024), Lebanon, New Hampshire
  - Cooper University Hospital (019-001), Camden, New Jersey
  - New Jersey Medical School Clinical Research Center (028-001), Newark, New Jersey
  - University of New Mexico Hospital (Site 213-008), Albuquerque, New Mexico
  - NYU Brooklyn (301-033), Brooklyn, New York
  - New York Presbyterian Queens (003-005), Flushing, New York
  - NYU Long Island (301-034), Mineola, New York
  - New York University Langone Health (301-013), New York, New York
  - NYC Health + Hospital Harlem (Site 003-003), New York, New York
  - Weill Cornell Clinical Research Unit (065-001), New York, New York
  - Mount Sinai Medical Center (Site 301-012), New York, New York
  - Lincoln Medical Center (Site 003-016), The Bronx, New York
  - James J. Peters VAMC (Site 023-003), The Bronx, New York
  - Duke University Hospital (Site 301-006), Durham, North Carolina
  - Wake Forest Baptist Health (Site 210-001), Winston-Salem, North Carolina
  - Cleveland Clinic Foundation (Site 207-001), Cleveland, Ohio
  - Oregon Health and Science University (208-003), Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center (Site 209-002), Hershey, Pennsylvania
  - Rhode Island Hospital (Site 080-036), Providence, Rhode Island
  - The Miriam Hospital (Site 080-039), Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center (074-015), Charleston, South Carolina
  - Medical University of South Carolina (Site 210-002), Charleston, South Carolina
  - Vanderbilt University Medical Center (Site 212-001), Nashville, Tennessee
  - Hendrick Medical Center (Site 080-014), Abilene, Texas
  - CHRISTUS Spohn Shoreline Hospital (080-001), Corpus Christi, Texas
  - Parkland Health and Hospital Systems (084-002), Dallas, Texas
  - Baylor, Scott and White Health (301-003), Dallas, Texas
  - UT Southwestern Medical Center (084-001), Dallas, Texas
  - Houston Methodist Research Institute (Site 301-028), Houston, Texas
  - University of Texas Health Science Center (Site 203-006), Houston, Texas
  - UT Health San Antonio (Site 009-022), San Antonio, Texas
  - Intermountain Medical Center (Site 211-001), Murray, Utah
  - University of Utah Hospital (211-002), Salt Lake City, Utah
  - Salem VA Medical Center (Site 074-014), Salem, Virginia
  - Harborview Medical Center (208-001), Seattle, Washington
  - Providence (Sacred Heart) (213-004), Spokane, Washington
  - West Virginia University Medicine (Site 301-023), Morgantown, West Virginia
  - William S. Middleton Memorial Veterans Hospital (074-030), Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital (052-001), Milwaukee, Wisconsin
- Australia (6):
  - St. Vincent's Hospital (Site 612-002), Sydney, New South Wales
  - Westmead Hospital (Site 612-058), Westmead, New South Wales
  - Royal Brisbane and Women's Hospital (612-055), Brisbane, Queensland
  - Monash Health (612-009), Clayton, Victoria
  - Austin Health (612-020), Heidelberg, Victoria
  - The Alfred Hospital (612-017), Melbourne, Victoria
- Denmark (8):
  - Odense University Hospital (625-004), Odense, C
  - Aalborg Hospital (Site 625-005), Aalborg
  - Aarhus Universitetshospital, Skejby (Site 625-002), Aarhus
  - Rigshospitalet, CHIP (Site 625-006), Copenhagen
  - Bispebjerg Hospital (Site 625-013), Copenhagen
  - Herlev/Gentofte Hospital (Site 625-012, Hellerup
  - Nordsjællands Hospital, Hillerød (Site 625-009), Hillerød
  - Hvidovre University Hospital, Department of Infectious Diseases (Site 625-001), Hvidovre
- Hôpital Saint André (Site 631-041), Bordeaux, France
- AIDS and Clinical Immunology Research Center (627-201), Tbilisi, Georgia
- Klinik I für Innere Medizin der Universität zu Köln (622-008), Cologne, Germany
- Greece (4):
  - 1st Respiratory Medicine Department, Athens University Medical School (635-015), Athens, Attica
  - 3rd Dept of Medicine, Medical School, NKUA (635-022), Athens, Attica
  - Attikon University General Hospital (Site 635-009), Athens, Attica
  - Democritus University of Thrace (635-021), Alexandroupoli, Evros
- Chennai Antiviral Research and Treatment Clinical Research Site (Site 612-402), Chennai, Tamil Nadu, India
- St Vincent's University Hospital (Site 634-103), Dublin, Ireland
- Institute of Human Virology-Nigeria (IHVN) (612-601), Abuja, Federal Capital Territory, Nigeria
- Wojewodzki Szpital Zakazny (Site 625-302), Warsaw, Poland
- Tan Tock Seng Hospital (Site 612-201), Singapore, Singapore
- South Korea (5):
  - Seoul National University Bundang Hospital (612-904), Seongnam
  - National Medical Center (612-905), Seoul
  - Asan Medical Center (612-901), Seoul
  - Seoul St. Mary's Hospital (Site 612-903), Seoul
  - Chung-Ang University Hospital (612-902), Seoul
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol (626-003), Badalona, Barcelona
  - Hospital del Mar (626-025), Barcelona
  - Hospital Universitari Vall d'Hebron (626-033), Barcelona
  - Hospital Clinic de Barcelona (626-004), Barcelona
  - Hospital Universitario La Paz (Site 626-012), Madrid
- Karolinska University Hospital, Solna (Site 625-206), Stockholm, Sweden
- University Hospital Basel (636-004), Basel, Switzerland
- Thailand (3):
  - Siriraj Hospital (613-002), Bangkok Noi, Bangkok
  - Chulalongkorn University and The HIV-NAT (Site 613-001), Bangkok
  - Khon Kaen University, Srinagarind Hospital (613-003), Khon Kaen
- Ukraine (3):
  - Central City Clinical Hospital of Ivano-Frankivsk City Council (627-302), Ivano-Frankivsk
  - Treatment and Diagnostic Center ADONIS Plus (627-304), Kyiv
  - Hospital #1 of Zhytomyr City Council (627-303), Zhytomyr
- University Hospital Plymouth NHS Trust (Site 634-014), Plymouth, Devon, United Kingdom